CLINICAL TRIAL: NCT02779530
Title: Evaluation of CYP4A11 and CYP4F2 Gene Variants as Makers in Edema and Elevated Blood Pressure Occurrence After Nonsteroidal Anti-inflammatory (NSAID) Use
Brief Title: CYP4A11 and CYP4F2 Gene Variants as Makers of Cardiovascular Adverse Events of Non-steroidal Anti-inflammatory Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eduardo Barbosa Coelho (Other)
Responsible Party: Sponsor-Investigator, Eduardo Barbosa Coelho, Associate Professor Nephrology Division - Internal Medicine Dept. Ribeirão Preto Medical School University of São Paulo, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Screening
Other Study IDs: U1111-1131-8461
Record Dates: First submitted 2016-05-17; First posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac (Experimental)
  Interventions: Drug: Diclofenac
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Diclofenac — 50 mg po, b.i.d for 6 days
  Arms: Diclofenac
Other: Placebo — Placebo po, b.i.d. for 6 days
  Arms: Placebo

SUMMARY:
Randomized, double-blinded, cross-over and placebo controlled clinical trial to evaluate the association between genetic polymorphism of CYP4F2 with cardiovascular adverse effects of non-steroidal anti-inflammatory drugs (NSAIDs). Two groups were included according the CYP4F2 V433M genetic polymorphism (control - MM, N=7 vs. VV or VM variants, N=13). According the sample size planned, a mean difference of total body water delta between groups (control vs. polymorphic) of at least allow 10% could be observed.

ELIGIBILITY:
Inclusion Criteria: Healthy volunteers 18-65 years-old -

Exclusion Criteria: Use of drugs and without clinical history of adverse effects of NSAIDS

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Edema | after 6 days of diclofenac and placebo
  Presence of edema, measured by the estimative of total body water (deuterium oxide dilution technique). The measurements will be done in the end of 6 days of use of placebo and diclofenac, and the delta between diclofenac and placebo will be used as endpoint

SECONDARY OUTCOMES:
Blood Pressure | after 6 days of diclofenac and placebo
  Variation (delta) of 24h diastolic blood pressure between placebo and diclofenac phases, measured by ambulatory blood pressure monitoring (ABPM)

CONTACTS AND LOCATIONS:
Locations (1):
- Unidade de Pesquisa Clínica HCRP-USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No